CLINICAL TRIAL: NCT04115332
Title: 精神科受暴護理人員復原力與心理健康之成效-以生理回饋訓練為介入措施 The Effects of Resilience and Mental Health of Abused Psychiatric Nurses: An Intervention With Biofeedback Training
Brief Title: The Effects of Resilience and Mental Health of Abused Psychiatric Nurses: An Intervention With Biofeedback Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: KMUHIRB-E(II)-20170101
Record Dates: First submitted 2019-10-01; First posted 2019-10-04 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2017-04

CONDITIONS: Psychiatric Nurses, Workplace Violence, Biofeedback Training, and Resilience
Keywords: psychiatric nurses; workplace violence; resilience; biofeedback training; physiological indicators

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional (Experimental): EEG Recording The one-channel EEG sensor was recorded from Cz with linked-ear reference based on the International 10-20 system. EEG signals were recorded using BioGraph Infiniti software (Version 6.0.4, n.d.) with a band-pass between 1-30 Hz. The sample rate was 256 Hz with 60-Hz notch filters, and the electrode impedances were lower than 5 kΩ.
  A lead II electrocardiogram (ECG) was collected for 5 minutes at baseline using the ProComp InfinitiTM system (Thought Technology Ltd., Montreal, Canada), which was installed on a laptop. A sampling rate of 2,048/second was set in order to acquire real-time interbeat intervals.
  Interventions: Biological: bio-feedback training

INTERVENTIONS:
Biological: bio-feedback training — The aim of this study was to explore the abused PW nurses who receiving bio-feedback training as an intervention improve, and change of physiological indicators before and after intervention (3 months later), which included Respiratory Rate (RR), skin conduction (SC), heart rate variability (HRV), and resilience.

SUMMARY:
The investigators provide biofeedback training to assist the abused PW nurses to reduce WPV-related stress and achieve better resilience and mental health. The research project will assess the participants' physiological indices prior to the intervention as well as their levels of resilience and mental status.

DETAILED DESCRIPTION:
This was a quasi-experimental study, structured questionnaires of Resilience Score, The Center for Epidemiologic Studies Depression (CES-D) and Occupational Stress Indicator-2 were used in this study before and three months after intervention. A total of 112 abused psychiatric nurses were randomly assigned to 3 groups. The biofeedback group (n=40) received the biofeedback training and the self-training group received video relaxation training by Line (n=44). The control group (n=28) did not receive any intervention.

Biofeedback training is an effective intervention to enhance abused PW nurses' resilience and lower their depressive symptoms. Video relaxation self-training is also an effective way to strengthen abused psychiatric nurses' resilience.

ELIGIBILITY:
Inclusion Criteria:

* abused psychiatric ward (PW) nurses

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2017-07-08 (Actual); Primary Completion 2017-10-08 (Actual); Study Completion 2017-10-08 (Actual)

PRIMARY OUTCOMES:
The Center for Epidemiologic Studies Depression | 15 minutes
  The Chinese version Center for Epidemiologic Studies Depression was developed with a Cronbach's alpha of 0_86, and it was used as the screening measure of depressive tendency in this study. The cut-off point of the scale is of greater than or equal to 15 on the CES-D score.
The Resilience | 15 minutes
  The Resilience Scale was developed by Friborg et al. (2006) and the Chinese version was established by Wang and Chen with satisfactory validity and reliability. The 29-item scale measures intrapersonal and interpersonal protective resources that may facilitate an individual's adaptability to and tolerance for stress and adverse life events. The scale comprises five components, including personal strength, social competence, structured style, family cohesion, and social resources. The total scores of the RS range from 29 to 203, with higher scores indicating a higher level of resilience.

SECONDARY OUTCOMES:
EEG | 5 minutes
  The one-channel EEG sensor was recorded from Cz with linked-ear reference based on the International 10-20 system. EEG signals were recorded using BioGraph Infiniti software (Version 6.0.4, n.d.) with a band-pass between 1-30 Hz.
Heart rate | 5 minutes
  electrocardiogram (ECG) was collected for 5 minutes at baseline using the ProComp InfinitiTM system (Thought Technology Ltd., Montreal, Canada), which was installed on a laptop. A sampling rate of 2,048/second was set in order to acquire real-time interbeat intervals.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Taiwan